CLINICAL TRIAL: NCT02570009
Title: Weight Loss for Couples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Amy Gorin, Associate Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HL125157
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Overweight; Obesity
Keywords: couples; weight loss treatment; home environment
MeSH Terms: conditions — Overweight; Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- TEAMS (Active Comparator)
  Interventions: Behavioral: TEAMS (Talking about Eating, Activity, Mutual Support)
- TEAMS+ (Active Comparator)
  Interventions: Behavioral: TEAMS (Talking about Eating, Activity, Mutual Support); Behavioral: Need Support Training

INTERVENTIONS:
Behavioral: TEAMS (Talking about Eating, Activity, Mutual Support)
Behavioral: Need Support Training
  Arms: TEAMS+

SUMMARY:
Obesity risk is shared within married couples yet most existing weight loss programs focus on individuals and not the marital dyad. This project will test the effects of a couples weight loss program that teaches spouses how to provide each other with autonomy support and create an interpersonal environment that promotes sustained behavior change.

ELIGIBILITY:
Inclusion Criteria:

18-70 years old interested in receiving free weight loss treatment with their spouse have a body mass index (BMI) between 25 and 45 kg/m2. Individuals who respond to the advertisement will be screened for eligibility by phone. Eligibility will be limited to married/cohabitating couples (n=64) in which each spouse is 18-70 years old with a BMI between 25-45 kg/m2.

Exclusion Criteria:

currently in a weight loss program, dieting, or taking medications that might affect weight participated in a weight loss program in the past year have lost > 10% of body weight during past 6 months are currently participating in any other research study that may interfere with this study are pregnant, lactating, < 6 months postpartum, or plan to become pregnant during the study have undergone cancer treatment within the past year, not including skin cancer treatment have substance abuse, dependence, average more than 14 drinks per week, or are currently being treated for alcohol or substance abuse have a heart condition, chest pain during periods of activity or rest, or loss of consciousness report uncontrolled hypertension, history of coronary heart disease, stroke, peripheral arterial disease or have a blood pressure ≥160/100 mmHG as measured by study staff at baseline report chronic gastrointestinal disease endorse having hepatitis B or C, cirrhosis, or HIV; or report a significant psychiatric illness that may interfere with completion of the study deemed by study staff to be unlikely to adhere to study protocol (e.g. moving in the next 12 months).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Weight loss | One year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

REFERENCES:
- [Derived] Gorin AA, Leahey TM, Cornelius T, Bourgea K, Powers TA. Self-control and grit: associations with weight management and healthy habits. J Behav Med. 2024 Feb;47(1):160-167. doi: 10.1007/s10865-023-00431-9. Epub 2023 Jul 13. PMID 37440156
- [Derived] Denes A, Crowley JP, Ponivas ALP, Cornelius T, Allred RJ, Gettens KM, Powers TA, Gorin AA. Evidence of the Associations between Individual and Partner Autonomy Support and Physiological Stress in the Context of Conversations about Weight among Couples Who are Overweight or Obese during a 6-Month Intervention. Health Commun. 2022 Jul;37(8):1013-1021. doi: 10.1080/10410236.2021.1880685. Epub 2021 Feb 9. PMID 33563035
- [Derived] Gorin AA, Powers TA, Gettens K, Cornelius T, Koestner R, Mobley AR, Pescatello L, Medina TH. Project TEAMS (Talking about Eating, Activity, and Mutual Support): a randomized controlled trial of a theory-based weight loss program for couples. BMC Public Health. 2017 Sep 29;17(1):749. doi: 10.1186/s12889-017-4732-7. PMID 28962602